CLINICAL TRIAL: NCT04113889
Title: Effects of Triple Drug Cocktail Therapy on Metabolic, Endocrine Alterations and Perceived Stress Response in Patients With PCOS: A Double Blind Randomized Clinical Trial
Brief Title: Effects of Triple Drug Cocktail Therapy on Metabolic, Endocrine Alterations and Perceived Stress in Patients With Poly Cystic Ovary Syndrome
Acronym: PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Mohsin Shah, Associate Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASRB001062/ET/IBMS
Record Dates: First submitted 2019-09-26; First posted 2019-10-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: PCOS
Keywords: PCOS; Acetyl-L-Carnitine
MeSH Terms: interventions — Metformin; Pioglitazone; Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination therapy group (Active Comparator): Arm 1: Metformin (1000 mg daily), Pioglitazone (30 mg daily), Acetyl-L-carnitine (3 gm daily)
  Interventions: Drug: Metformin (1000 mg daily), Pioglitazone (30 mg daily), Acetyl-L-carnitine (3 gm daily)
- Standard therapy group (Placebo Comparator): Arm 2: Metformin (1000 mg daily), Pioglitazone (30 mg daily), Placebo
  Interventions: Drug: Metformin, pioglitazone and placebo

INTERVENTIONS:
Drug: Metformin (1000 mg daily), Pioglitazone (30 mg daily), Acetyl-L-carnitine (3 gm daily) — 72 patients with PCOS receiving metformin, pioglitazone and Acetyl L-Carnitine 500 mg, 15 mg and 1.5 gm BD daily respectively.
  Other Names: Zolid plus and Acetyl-L-carnitine
  Arms: Combination therapy group
Drug: Metformin, pioglitazone and placebo — 72 patients with PCOS receiving metformin, pioglitazone and placebo 500 mg, 15 mg and placebo BD daily respectively.
  Other Names: Zolid plus and placebo
  Arms: Standard therapy group

SUMMARY:
The investigators aim is to conduct a double blind randomized clinical trial, to study the effects of triple drug cocktail (metformin, pioglitazone and acetyl L-Carnitine) therapy on metabolic, endocrine alterations and perceived stress response in patients with Polycystic Ovary Syndrome (PCOS). Women diagnosed with PCOS, using criteria proposed in November 2015, by the American Association of Clinical Endocrinologists (AACE), American College of Endocrinology (ACE), and Androgen Excess and PCOS Society (AES) for PCOS should include two of the following three criteria: chronic an ovulation, hyperandrogenism (clinical/biologic), and polycystic ovaries. The investigators propose that PCOS women may have altered metabolic, endocrine levels and increased perceived stress response and combination therapy may have beneficial influences on these parameters in women diagnosed with PCOS.

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome (PCOS) is an endocrinopathy which affects 5-10% of reproductive age women (1). The three main features of the syndrome are polycystic ovaries, high levels of androgen in blood and chronic an-ovulation/oligo-an ovulation (2). Women with PCOS have a greater risk of developing hyperinsulinemia and insulin resistance (3). PCOS may lead to insulin resistance and dyslipidemia (3). Recent long-term follow up studies of the syndrome have shown that women suffering from the syndrome have hyperlipidemia and enhanced risk of cardiovascular diseases (3).

Recent evidence has demonstrated that anti-inflammatory drug treatments ameliorate insulin resistance. Metformin belongs to a family of drugs called the biguanides, currently used as an antihyperglycemic drug for treatment of type II diabetes mellitus (4). Around 15 years ago it was reported for the first time that use of metformin in PCOS effectively reduced insulin resistance (4). Increasing evidence has shown the importance of metformin not only in hyperinsulinemic patients but also in PCOS resolving several other issues like menstrual cycles, fertility, hormonal imbalance and metabolic syndromes (4). Pioglitazone is a drug from class thiazolidinedione (TZD) with hypoglycemic (anti-hyperglycemic, anti-diabetic) action in the management of type 2 diabetes (5). Recent studies have shown that pioglitazone may be considered a new treatment option for patients with PCOS, since it is able to restore normal menstrual cycle and have improved ovulation (6). Recent randomized placebo controlled clinical trials have also shown that it is associated with good serum lipid profile levels (7).

Acetyl L-Carnitine is an isomer synthesized by two amino acids lysine and methionin mainly distributed among skeletal and cardiac muscles in mammals (8, 9). Acetyl L-Carnitine is involved in fatty acid oxidation by transporting long chain fatty acids into mitochondria for oxidation to produce metabolic energy and have effects on oxidative metabolism of glucose in tissues (9). Acetyl L-Carnitine is known to regulate energy production (10). Studies have shown that patients treated with acetyl L-Carnitine have improved ovulation and pregnancy rates and is well tolerated by the patients (8). PCOS patients have shown reduced adiponectin levels associated with insulin resistance states and type 2 diabetes mellitus and treatment with L-Carnitine has shown reduced blood glucose levels, increased insulin sensitivity and also improved adiponectin levels, which can be attributed to L-carnitine-induced increase in beta-oxidation of fatty acids and basal metabolic rates (11).

PCOS is a systemic condition, an endocrinopathy whose etiology is still not understood. Correct treatment regimens of PCOS will not only improve menstrual cycles of the patients but will also improve the metabolic or endocrine parameters (2). PCOS sufferers are also known to have increased perceived stress response which will be considered in the study. Little evidences are available on combination therapy for treatment of PCOS patients. The aim of this study is to come up with a better treatment option to ameliorate the signs and symptoms associated with the disease.

Study objectives:

To find the effects of triple drug cocktail therapy (metformin, pioglitazone and acetyl L-Carnitine) on metabolic, endocrine alterations and perceived stress response in patients with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naive PCOS women having age from 14-45 years with scanty or no menstruation, hirsutism and elevated serum androgen levels, will be diagnosed on the basis of AES (Androgen access society) guidelines 2006 according to which when two of the following criteria are present patient will be said to have the syndrome
2. Hirsutism or hyperandrogenism
3. Oligo or an-ovulation and or polycystic ovaries -

Exclusion Criteria:

1. Women with previous history of Cushing syndrome
2. Thyroid disorders
3. Hyperprolactinemia
4. Ovarian tumors
5. Congenital adrenal hyperplasia androgen-producing tumors,
6. History of seizures
7. Patients on warfarin, Coumadin and Sintrom because of drug interaction with acetyl-L-Carnitine,
8. Pregnancy or using contraceptive medications,
9. Patients on hormonal therapy that alters the biochemical or hormonal profile

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 3 months
  PCOS associated insulin resistance and hyperinsulinemia through HOMA-IR
Hypoadiponectinemia | 3 months
  PCOS associated Hypoadiponectinemia. Measurement of adiponectin level through ELISA
Ovary volume | 3 months
  Polycystic ovaries volume measurement by abdominal ultrasound
Stress response | 3 months
  Perceived stress response and profile of mood stress by structured questionnaire

SECONDARY OUTCOMES:
Body fat analysis | 3 months
  Body fats measurement through measurement scale
Hirsutism | 3 months
  Hirsutism score
Menstrual irregularities | 3 months
  Oligo/anovulation
Androgenic Alopecia | 3 months
  Hair on head area
Pregnancy | 3 months
  Fertility/infertility

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Shah, PhD, Principal Investigator — Department of Physiology, Khyber Medical University, Peshawar Pakistan
Locations (1):
- Gynecology and Obstetric, Hayatabad Medical Complex, Peshawar, Khyber Pukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nestler JE, Stovall D, Akhter N, Iuorno MJ, Jakubowicz DJ. Strategies for the use of insulin-sensitizing drugs to treat infertility in women with polycystic ovary syndrome. Fertil Steril. 2002 Feb;77(2):209-15. doi: 10.1016/s0015-0282(01)02963-6. PMID 11821072
- [Background] Elkind-Hirsch K, Marrioneaux O, Bhushan M, Vernor D, Bhushan R. Comparison of single and combined treatment with exenatide and metformin on menstrual cyclicity in overweight women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Jul;93(7):2670-8. doi: 10.1210/jc.2008-0115. Epub 2008 May 6. PMID 18460557
- [Background] Glintborg D, Andersen M, Hagen C, Heickendorff L, Hermann AP. Association of pioglitazone treatment with decreased bone mineral density in obese premenopausal patients with polycystic ovary syndrome: a randomized, placebo-controlled trial. J Clin Endocrinol Metab. 2008 May;93(5):1696-701. doi: 10.1210/jc.2007-2249. Epub 2008 Feb 19. PMID 18285411
- [Background] Xu Y, Wu Y, Huang Q. Comparison of the effect between pioglitazone and metformin in treating patients with PCOS:a meta-analysis. Arch Gynecol Obstet. 2017 Oct;296(4):661-677. doi: 10.1007/s00404-017-4480-z. Epub 2017 Aug 2. PMID 28770353
- [Background] Ismail AM, Hamed AH, Saso S, Thabet HH. Adding L-carnitine to clomiphene resistant PCOS women improves the quality of ovulation and the pregnancy rate. A randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2014 Sep;180:148-52. doi: 10.1016/j.ejogrb.2014.06.008. Epub 2014 Jun 23. PMID 25015747
- [Background] Rajasekar P, Anuradha CV. Effect of L-carnitine on skeletal muscle lipids and oxidative stress in rats fed high-fructose diet. Exp Diabetes Res. 2007;2007:72741. doi: 10.1155/2007/72741. PMID 17641743
- [Background] Bernard A, Rigault C, Mazue F, Le Borgne F, Demarquoy J. L-carnitine supplementation and physical exercise restore age-associated decline in some mitochondrial functions in the rat. J Gerontol A Biol Sci Med Sci. 2008 Oct;63(10):1027-33. doi: 10.1093/gerona/63.10.1027. PMID 18948552
- [Derived] Tauqir S, Israr M, Rauf B, Malik MO, Habib SH, Shah FA, Usman M, Raza MA, Shah I, Badshah H, Ehtesham E, Shah M. Acetyl-L-Carnitine Ameliorates Metabolic and Endocrine Alterations in Women with PCOS: A Double-Blind Randomized Clinical Trial. Adv Ther. 2021 Jul;38(7):3842-3856. doi: 10.1007/s12325-021-01789-5. Epub 2021 May 28. PMID 34047916